CLINICAL TRIAL: NCT01648660
Title: Long Term Effects of Lutein/Zeaxanthin and Omega-3- Supplementation on Optical Density of AMD Patients for Two More Years (LUTEGA 2)
Brief Title: Long Term Effects of Lutein/Zeaxanthin and Omega-3- Supplementation for Two More Years (LUTEGA 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Jens Dawczynski, Prof. Dr. med. Jens Dawczynski, University of Leipzig
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2032- 06/07
Record Dates: First submitted 2012-07-19; First posted 2012-07-24 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Age Related Maculopathy
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein; Zeaxanthins; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- D2x - D1x (Active Comparator): Cross Over from double dosage to single dosage:
  daily supplementation with 10mg Lutein, 1mg Zeaxanthin, 255 mg Omega-3-FAabout two years after one year with 20mg Lutein, 2mg Zeaxanthin, 510 mg Omega-3-FA
  Interventions: Dietary Supplement: Lutein/ Zeaxanthin + Omega- 3- Fatty Acids
- D1x - D2x (Active Comparator): Cross Over from double dosage to single dosage:
  daily supplementation with 20mg Lutein, 2mg Zeaxanthin, 510 mg Omega-3-FA about two years after one year with 10mg Lutein, 1mg Zeaxanthin, 255 mg Omega-3-FA
  Interventions: Dietary Supplement: Lutein/ Zeaxanthin + Omega- 3- Fatty Acids
- D1x - D1x (Active Comparator): single dosage: daily supplementation about two years after one year with 10mg Lutein, 1mg Zeaxanthin, 255 mg Omega-3-FA (dosage remains existing)
  Interventions: Dietary Supplement: Lutein/ Zeaxanthin + Omega- 3- Fatty Acids

INTERVENTIONS:
Dietary Supplement: Lutein/ Zeaxanthin + Omega- 3- Fatty Acids — capsule with Lutein, Zeaxanthin, Omega-3-FA for two years

SUMMARY:
The primary objective of LUTEGA 2 is it to determine the long term effect (about 2 more years after LUTEGA 1, NCT00763659) of the supplementation with a fixed combination of lutein/zeaxanthin and omega-3- fatty acids in two different dosages on the optical density (OD) of macular pigment in patients with non- exudative age related maculopathy. The dosage groups are crossed after LUTEGA 1.

DETAILED DESCRIPTION:
The LUTEGA 2 is a cross-over- study and the continue of LUTEGA 1. After one year of supplementation in randomized, placebo- controlled, double blind study (LUTEGA 1), the treatment arms are unblind to cross over the different dosage groups.

The measurement of optical density of macular pigment (MPOD) uses the 1- wavelength reflection method recording reflection images at 480 nm by a fundus camera. The patients are followed up over two years in eight more visits (every three months) In addition to the MPOD- measurement each examination includes standardized visual acuity test (ETDRS), amsler- grid, slit lamp biomicroscopy, fundus photography (color and autofluorescence) and a blood sample (every six months).

ELIGIBILITY:
Inclusion Criteria:

* All non- exudative forms of age related maculopathy

Exclusion Criteria:

* Exudative age related maculopathy
* decrease opacity of ocular media

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Optical density of macular pigment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Strobel, MD, Study Director — University Hospital Jena; Jens Dawczynski, MD, Principal Investigator — University of Leipzig